CLINICAL TRIAL: NCT00321464
Title: A Randomized, Double-Blind, Multicenter Study of Denosumab Compared With Zoledronic Acid (Zometa®) in the Treatment of Bone Metastases in Subjects With Advanced Breast Cancer
Brief Title: A Study Comparing Denosumab vs. Zoledronic Acid for the Treatment of Bone Metastases in Breast Cancer Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20050136
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Bone Metastases
Keywords: Fractures; Compressions; Bisphosphonates; Bone metastases; Breast cancer; Skeletal; Radiation; Surgery to Bone
MeSH Terms: conditions — Fractures, Bone; Breast Neoplasms | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zoledronic acid (Active Comparator)
  Interventions: Drug: Zoledronic Acid
- denosumab (Experimental)
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — Q4W 120 mg denosumab SC injection and 4 mg zoledronic acid (Zometa) placebo IV over a minimum of 15 minutes
  Arms: denosumab
Drug: Zoledronic Acid — Q4W 4 mg zoledronic acid IV over minimum 15 minutes and 120 mg denosumab placebo SC
  Other Names: Zometa
  Arms: zoledronic acid

SUMMARY:
The purpose of this study is to determine if denosumab is non-inferior to zoledronic acid in the treatment of bone metastases in subjects with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults with histologically or cytologically confirmed breast adenocarcinoma
* radiographic evidence of at least one bone mets
* Easter Cooperative Oncology Group status of 0, 1 or 2;
* adequate organ function

Exclusion Criteria:

* Current or prior IV bisphosphonate administration
* current or prior oral bisphosphonates for bone mets
* life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2049 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2009-07-20 (Actual); Study Completion 2012-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Cleeland CS, Body JJ, Stopeck A, von Moos R, Fallowfield L, Mathias SD, Patrick DL, Clemons M, Tonkin K, Masuda N, Lipton A, de Boer R, Salvagni S, Oliveira CT, Qian Y, Jiang Q, Dansey R, Braun A, Chung K. Pain outcomes in patients with advanced breast cancer and bone metastases: results from a randomized, double-blind study of denosumab and zoledronic acid. Cancer. 2013 Feb 15;119(4):832-8. doi: 10.1002/cncr.27789. Epub 2012 Sep 5. PMID 22951813
- [Background] Martin M, Bell R, Bourgeois H, Brufsky A, Diel I, Eniu A, Fallowfield L, Fujiwara Y, Jassem J, Paterson AH, Ritchie D, Steger GG, Stopeck A, Vogel C, Fan M, Jiang Q, Chung K, Dansey R, Braun A. Bone-related complications and quality of life in advanced breast cancer: results from a randomized phase III trial of denosumab versus zoledronic acid. Clin Cancer Res. 2012 Sep 1;18(17):4841-9. doi: 10.1158/1078-0432.CCR-11-3310. Epub 2012 Aug 14. PMID 22893628
- [Background] Stopeck AT, Lipton A, Body JJ, Steger GG, Tonkin K, de Boer RH, Lichinitser M, Fujiwara Y, Yardley DA, Viniegra M, Fan M, Jiang Q, Dansey R, Jun S, Braun A. Denosumab compared with zoledronic acid for the treatment of bone metastases in patients with advanced breast cancer: a randomized, double-blind study. J Clin Oncol. 2010 Dec 10;28(35):5132-9. doi: 10.1200/JCO.2010.29.7101. Epub 2010 Nov 8. PMID 21060033
- [Derived] Stopeck AT, Fizazi K, Body JJ, Brown JE, Carducci M, Diel I, Fujiwara Y, Martin M, Paterson A, Tonkin K, Shore N, Sieber P, Kueppers F, Karsh L, Yardley D, Wang H, Maniar T, Arellano J, Braun A. Safety of long-term denosumab therapy: results from the open label extension phase of two phase 3 studies in patients with metastatic breast and prostate cancer. Support Care Cancer. 2016 Jan;24(1):447-455. doi: 10.1007/s00520-015-2904-5. Epub 2015 Sep 3. PMID 26335402
- [Derived] Body JJ, Bone HG, de Boer RH, Stopeck A, Van Poznak C, Damiao R, Fizazi K, Henry DH, Ibrahim T, Lipton A, Saad F, Shore N, Takano T, Shaywitz AJ, Wang H, Bracco OL, Braun A, Kostenuik PJ. Hypocalcaemia in patients with metastatic bone disease treated with denosumab. Eur J Cancer. 2015 Sep;51(13):1812-21. doi: 10.1016/j.ejca.2015.05.016. Epub 2015 Jun 17. PMID 26093811
- [Derived] Diel IJ, Body JJ, Stopeck AT, Vadhan-Raj S, Spencer A, Steger G, von Moos R, Goldwasser F, Feng A, Braun A. The role of denosumab in the prevention of hypercalcaemia of malignancy in cancer patients with metastatic bone disease. Eur J Cancer. 2015 Jul;51(11):1467-75. doi: 10.1016/j.ejca.2015.04.017. Epub 2015 May 11. PMID 25976743
- [Derived] von Moos R, Body JJ, Egerdie B, Stopeck A, Brown JE, Damyanov D, Fallowfield LJ, Marx G, Cleeland CS, Patrick DL, Palazzo FG, Qian Y, Braun A, Chung K. Pain and health-related quality of life in patients with advanced solid tumours and bone metastases: integrated results from three randomized, double-blind studies of denosumab and zoledronic acid. Support Care Cancer. 2013 Dec;21(12):3497-507. doi: 10.1007/s00520-013-1932-2. Epub 2013 Aug 22. PMID 23975226
- [Derived] Lipton A, Fizazi K, Stopeck AT, Henry DH, Brown JE, Yardley DA, Richardson GE, Siena S, Maroto P, Clemens M, Bilynskyy B, Charu V, Beuzeboc P, Rader M, Viniegra M, Saad F, Ke C, Braun A, Jun S. Superiority of denosumab to zoledronic acid for prevention of skeletal-related events: a combined analysis of 3 pivotal, randomised, phase 3 trials. Eur J Cancer. 2012 Nov;48(16):3082-92. doi: 10.1016/j.ejca.2012.08.002. Epub 2012 Sep 10. PMID 22975218
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 27 April 2006 through 31 December 2007
Pre-assignment Details: 2049 patients were enrolled in the study, but 3 patients were excluded from all analyses because properly documented informed consent was not obtained.
Groups:
- Zoledronic Acid: Zoledronic acid 4 mg by intravenous injection with subcutaneous denosumab placebo once every 4 weeks
- Denosumab: Denomsumab 120 mg subcutaneously with intravenous zoledronic acid placebo once every 4 weeks
Period: Overall Study
Arm/Group | Zoledronic Acid | Denosumab
Started | 1020 | 1026
Received Investigational Product | 1014 | 1019
Completed | 461 | 468
Not Completed | 559 | 558
Not completed — Death | 169 | 174
Not completed — Disease progression | 124 | 124
Not completed — Withdrawal by Subject | 117 | 118
Not completed — Participant request | 57 | 61
Not completed — Adverse Event | 43 | 28
Not completed — Physician Decision | 15 | 14
Not completed — Noncompliance | 4 | 10
Not completed — Lost to Follow-up | 7 | 8
Not completed — Protocol deviation | 0 | 2
Not completed — Ineligibility determined | 2 | 1
Not completed — Other | 21 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Denosumab | Total
Number analyzed (Participants) | 1020 | 1026 | 2046
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (11.6) | 56.8 (11.5) | 56.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1011 | 1018 | 2029
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 813 | 822 | 1635
  Black or African American | 25 | 26 | 51
  Hispanic or Latino | 59 | 59 | 118
  Asian | 37 | 32 | 69
  Japanese | 69 | 70 | 139
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Other | 16 | 16 | 32
Previous Skeletal-Related Event Stratification Factor [Number; unit: Participants]
  Yes | 373 | 378 | 751
  No | 647 | 648 | 1295
Prior Oral Bisphosphonate Use Stratification Factor [Number; unit: Participants]
  Yes | 38 | 42 | 80
  No | 982 | 984 | 1966
Current Chemotherapy Stratification Factor [Number; unit: Participants] — Defined as within 6 weeks before randomization
  Participants
    Yes | 408 | 410 | 818
    No | 612 | 616 | 1228
Japan Stratification Factor [Number; unit: Participants] — Participant located in Japan
  Participants
    Yes | 67 | 69 | 136
    No | 953 | 957 | 1910

OUTCOME MEASURES:

1. Primary Outcome: Time to First On-Study Skeletal Related Event (SRE) (Non-inferiority)
Description: Time to first on-study skeletal-related event (SRE) using a non-inferiority analysis. The median time to first skeletal-related event could not be estimated in one treatment arm, so the subject incidence is presented.
Time Frame: Up to 34 months
Population: Full Analysis Set, composed of all randomized participants.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 1020 | 1026
Participants | 372 | 315
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Non-Inferiority or Equivalence — A synthesis method was used for the non-inferiority test for the hypothesis that denosumab preserves at least 50% of the effect of zoledronic acid vs. placebo; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI [0.71 to 0.95] — Stratified by the randomization stratification factors (previous skeletal-related event, prior oral bisphosphonate use, current chemotherapy, and location in Japan)

2. Secondary Outcome: Time to First On-Study Skeletal-Related Event (Superiority)
Description: Time to first on-study skeletal-related event (SRE) using a superiority analysis. The median time to first skeletal-related event could not be estimated in one treatment arm, so the subject incidence is presented.
Time Frame: Up to 34 months
Population: Full Analysis Set, composed of all randomized participants.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 1020 | 1026
Participants | 372 | 315
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Superiority or Other; p = 0.010, Regression, Cox — P-value was adjusted for multiplicity according to a hierarchical testing strategy and Hochberg procedure; Hazard Ratio (HR) = 0.82, 95% CI [0.71 to 0.95] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to First and Subsequent On-Study Skeletal-Related Event
Description: Time to first and subsequent on-study skeletal-related event (SRE) using a multiple event analysis. To be considered a subsequent SRE, the event must occur at least 21 days after the previous SRE. This outcome measure utilizes multiple event times, was analyzed based on a proportional mean model, and is therefore more appropriately summarized by the cumulative number of events.
Time Frame: Up to 34 months
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Events
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 1020 | 1026
Events | 608 | 474
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Superiority or Other; p = 0.001, Anderson-Gill model — P-value was adjusted for multiplicity according to a hierarchical testing strategy and Hochberg procedure; Rate ratio = 0.77, 95% CI [0.66 to 0.89] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: up to 2 years 10 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  One subject who was randomized to zoledronic acid and received denosumab as the 1st investigational product was analyzed on the denosumab arm for safety analyses.
Arm/Group | Zoledronic Acid 4 mg Q4W | Denosumab 120 mg Q4W
Serious Adverse Events (participants affected / at risk) | 471/1013 | 453/1020
Other Adverse Events (participants affected / at risk) | 941/1013 | 924/1020
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4 mg Q4W (N=1013) | Denosumab 120 mg Q4W (N=1020)
Anaemia (Blood and lymphatic system disorders) | 32 | 27
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 22 | 17
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 6 | 6
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 14 | 16
Pancytopenia (Blood and lymphatic system disorders) | 2 | 5
Platelet disorder (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 12
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 3
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 4 | 1
Cardiac failure (Cardiac disorders) | 7 | 6
Cardiac failure acute (Cardiac disorders) | 0 | 3
Cardiac failure congestive (Cardiac disorders) | 5 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 4 | 6
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 2 | 1
Cardiopulmonary failure (Cardiac disorders) | 4 | 2
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Cytotoxic cardiomyopathy (Cardiac disorders) | 0 | 2
Left ventricular failure (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 2 | 3
Pericarditis (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 3
Endocrine disorder (Endocrine disorders) | 1 | 0
Amaurosis (Eye disorders) | 3 | 1
Cataract (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Exophthalmos (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 0 | 1
Macular oedema (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 2
Visual acuity reduced (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 14 | 15
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3
Ascites (Gastrointestinal disorders) | 5 | 10
Caecitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 5 | 3
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 16 | 19
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 3
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocele (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 3
Intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 23 | 21
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 31 | 31
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 14 | 12
Catheter site pain (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 2
Chest pain (General disorders) | 9 | 5
Chills (General disorders) | 2 | 3
Condition aggravated (General disorders) | 1 | 0
Crepitations (General disorders) | 1 | 0
Death (General disorders) | 1 | 2
Disease progression (General disorders) | 12 | 11
Drowning (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 5 | 15
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 15 | 20
Generalised oedema (General disorders) | 1 | 1
Impaired healing (General disorders) | 2 | 0
Implant expulsion (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 3
Multi-organ failure (General disorders) | 9 | 9
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 5 | 4
Organ failure (General disorders) | 1 | 0
Pain (General disorders) | 8 | 4
Performance status decreased (General disorders) | 2 | 0
Pyrexia (General disorders) | 26 | 21
Sudden death (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 2 | 2
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic congestion (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 16 | 24
Hepatic function abnormal (Hepatobiliary disorders) | 7 | 10
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatorenal failure (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 2
Jaundice (Hepatobiliary disorders) | 0 | 5
Liver disorder (Hepatobiliary disorders) | 3 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abdominal wall infection (Infections and infestations) | 1 | 0
Abscess jaw (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 1
Breast cellulitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2
Candida sepsis (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 3 | 3
Catheter sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 7
Clostridial infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2
Ear infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 3
Escherichia bacteraemia (Infections and infestations) | 3 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 0
Infection (Infections and infestations) | 2 | 2
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Mastitis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 3 | 0
Oral fungal infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 0
Periodontal infection (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 25 | 20
Pneumonia primary atypical (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 3
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 2
Septic shock (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Stenotrophomonas sepsis (Infections and infestations) | 2 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 9 | 7
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 12 | 11
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 4 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 2 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Incorrect route of drug administration (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation myelopathy (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Recall phenomenon (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 2
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Aspiration bronchial (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Blood culture positive (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 2 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 3
Hepatic enzyme increased (Investigations) | 1 | 2
International normalised ratio increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 0 | 2
Renal function test abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 1
White blood cell count abnormal (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 7 | 10
Cachexia (Metabolism and nutrition disorders) | 7 | 6
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 24 | 13
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 10 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 10
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 11 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 8
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 | 17
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 7
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Contralateral breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 6
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to biliary tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 46 | 47
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 | 20
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 6
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 9
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Paraneoplastic dermatomyositis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 2 | 0
Aphonia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Brain compression (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 5 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 2 | 1
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 10 | 8
Cranial nerve paralysis (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 2
Diplegia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 7
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 0 | 2
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 9 | 13
Hemiparesis (Nervous system disorders) | 2 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 6 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 2 | 2
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 2
Lethargy (Nervous system disorders) | 3 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 2
Meningism (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 4 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Phrenic nerve paralysis (Nervous system disorders) | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 3 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 8 | 6
Stupor (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 6
Transient ischaemic attack (Nervous system disorders) | 1 | 4
Tremor (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 6 | 3
Depression (Psychiatric disorders) | 1 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 2
Anuria (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 9 | 1
Renal failure acute (Renal and urinary disorders) | 6 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 2
Ovarian mass (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1
Urogenital prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 | 53
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 25 | 24
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 18 | 11
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 20 | 20
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Abdominal cavity drainage (Surgical and medical procedures) | 1 | 0
Arterial bypass operation (Surgical and medical procedures) | 0 | 1
Breast reconstruction (Surgical and medical procedures) | 0 | 1
Colostomy closure (Surgical and medical procedures) | 1 | 0
Mastectomy (Surgical and medical procedures) | 1 | 4
Oophorectomy (Surgical and medical procedures) | 0 | 1
Pleurodesis (Surgical and medical procedures) | 0 | 1
Radical hysterectomy (Surgical and medical procedures) | 0 | 1
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 0 | 1
Simple mastectomy (Surgical and medical procedures) | 1 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0
Cardiovascular insufficiency (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 8 | 4
Embolism (Vascular disorders) | 2 | 0
Endocrine hypertension (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Haemodynamic instability (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 3
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 8 | 5
Hypovolaemic shock (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lymphangiopathy (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 2 | 2
Thrombosis (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4 mg Q4W (N=1013) | Denosumab 120 mg Q4W (N=1020)
Anaemia (Blood and lymphatic system disorders) | 217 | 183
Leukopenia (Blood and lymphatic system disorders) | 72 | 78
Neutropenia (Blood and lymphatic system disorders) | 118 | 114
Thrombocytopenia (Blood and lymphatic system disorders) | 53 | 62
Abdominal pain (Gastrointestinal disorders) | 113 | 114
Abdominal pain upper (Gastrointestinal disorders) | 80 | 68
Constipation (Gastrointestinal disorders) | 203 | 175
Diarrhoea (Gastrointestinal disorders) | 198 | 223
Dyspepsia (Gastrointestinal disorders) | 73 | 52
Nausea (Gastrointestinal disorders) | 377 | 350
Stomatitis (Gastrointestinal disorders) | 70 | 90
Toothache (Gastrointestinal disorders) | 37 | 57
Vomiting (Gastrointestinal disorders) | 225 | 199
Asthenia (General disorders) | 192 | 187
Chest pain (General disorders) | 79 | 90
Chills (General disorders) | 56 | 26
Fatigue (General disorders) | 323 | 291
Mucosal inflammation (General disorders) | 60 | 68
Oedema peripheral (General disorders) | 146 | 172
Pain (General disorders) | 91 | 68
Pyrexia (General disorders) | 231 | 157
Influenza (Infections and infestations) | 54 | 57
Nasopharyngitis (Infections and infestations) | 94 | 83
Upper respiratory tract infection (Infections and infestations) | 58 | 55
Urinary tract infection (Infections and infestations) | 86 | 68
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 54 | 35
Rib fracture (Injury, poisoning and procedural complications) | 93 | 82
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 76 | 63
Aspartate aminotransferase increased (Investigations) | 53 | 35
Weight decreased (Investigations) | 92 | 78
Anorexia (Metabolism and nutrition disorders) | 171 | 176
Arthralgia (Musculoskeletal and connective tissue disorders) | 289 | 246
Back pain (Musculoskeletal and connective tissue disorders) | 256 | 238
Bone pain (Musculoskeletal and connective tissue disorders) | 233 | 181
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 77 | 81
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 147 | 147
Myalgia (Musculoskeletal and connective tissue disorders) | 106 | 82
Neck pain (Musculoskeletal and connective tissue disorders) | 71 | 64
Pain in extremity (Musculoskeletal and connective tissue disorders) | 221 | 199
Dizziness (Nervous system disorders) | 110 | 102
Headache (Nervous system disorders) | 210 | 193
Neuropathy peripheral (Nervous system disorders) | 71 | 71
Paraesthesia (Nervous system disorders) | 72 | 68
Peripheral sensory neuropathy (Nervous system disorders) | 51 | 50
Anxiety (Psychiatric disorders) | 73 | 74
Depression (Psychiatric disorders) | 85 | 71
Insomnia (Psychiatric disorders) | 136 | 123
Cough (Respiratory, thoracic and mediastinal disorders) | 179 | 171
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 173 | 197
Alopecia (Skin and subcutaneous tissue disorders) | 142 | 159
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 91 | 91
Pruritus (Skin and subcutaneous tissue disorders) | 66 | 57
Rash (Skin and subcutaneous tissue disorders) | 99 | 96
Hot flush (Vascular disorders) | 70 | 66
Hypertension (Vascular disorders) | 64 | 64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.